CLINICAL TRIAL: NCT04414332
Title: Registry of Angiovac Procedures In Detail Outcomes Database
Brief Title: Registry of Angiovac Procedures In Detail Outcomes Database-RAPID Registry
Acronym: RAPID
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John Moriarty, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: 2015-SEP-1 Amendment 5
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Venous Thromboembolic Disease; Deep Venous Thrombosis; Right Heart Pathology; Pulmonary Embolism
Keywords: inferior vena cava (IVC) clots; right atrial (RA) masses; pulmonary emboli (PE)
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection only — This registry is to capture high quality patient safety and effectiveness data on use of the Angiovac device for 3 separate, but overlapping conditions; a) Iliofemoral and Caval DVT, b) Right heart masses, and c) PE. The goal will be achieved by capturing a concise set of immediate and short-term functional and clinical outcome data for all patients who have the angiovac catheter deployed into the vascular system.

SUMMARY:
Venous thromboembolic disease is a significant cause of morbidity and mortality. The purpose of the RAPID registry is to collect information on the Angiovac procedure and Angiovac device used in the treatment of deep venous thrombosis (DVT), right heart pathology and pulmonary embolism.

DETAILED DESCRIPTION:
Venous thromboembolic disease is a significant cause of morbidity and mortality. Thrombolytic therapy has been shown to be a successful treatment modality, however its use is somewhat limited due to the known risk of hemorrhage (overall 22%, with up to 3% intracranial hemorrhage), and suggested risk of distal embolization where large mobile thrombi are encountered. In patients where either thrombolysis is contraindicated or unsuccessful and conventional therapies inadequate, bulk thrombectomy may be considered. Until recently this was primarily achieved with surgical thrombectomy; however the Angiovac device is posited to offer a minimally invasive alternative.

This registry will collect data on patients in whom the Angiovac device was placed into the body for management of inferior vena cava (IVC) clots, right atrial (RA) masses or pulmonary emboli (PE) will be included.

This registry is to capture high quality patient safety and effectiveness data on use of the Angiovac device for 3 separate, but overlapping conditions; a) Iliofemoral and Caval DVT, b) Right heart masses, and c) PE. The goal will be achieved by capturing a concise set of immediate and short-term functional and clinical outcome data for all patients who have the angiovac catheter deployed into the vascular system.

Any center performing Angiovac procedure and wishing to contribute patient data will be offered participation in the registry. These core sites will be required to submit the registry protocol for Institutional Review Board (IRB) review. Once documentation of IRB approval has been received, centers may transmit their data via secure REDCap (Research Electronic Data Capture) database in accordance with federal regulations in the Health Insurance Portability and Accountability Act (HIPAA

ELIGIBILITY:
Inclusion Criteria:

* All patients in whom the Angiovac device was placed into the body for removal of fresh, soft thrombi or emboli during extracorporeal bypass for up to 6 hours.

Exclusion Criteria:

* Angiovac device not deployed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ages 18 years and older in whom the Angiovac device was deployed.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Post procedure outcomes | Procedure and up to 24 hours post procedure
  to collect information on the Angiovac procedure and Angiovac device used in the treatment of deep venous thrombosis (DVT), right heart pathology and pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: John Moriarty, MD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: Yes
Share de-identified information regarding procedure specifics as per case report forms and procedure outcomes
Supporting Information: Study Protocol
Time Frame: as per individual contract

REFERENCES:
- [Derived] Moriarty JM, Liao M, Kim GHJ, Yang E, Desai K, Ranade M, Plotnik AN. Procedural outcomes associated with use of the AngioVac System for right heart thrombi: A safety report from RAPID registry data. Vasc Med. 2022 Jun;27(3):277-282. doi: 10.1177/1358863X211073974. Epub 2022 Feb 17. PMID 35176918